CLINICAL TRIAL: NCT03415061
Title: Does Intranasal Insulin Administration Reduce the Incidence of Cognitive Dysfunction After Cardiac Surgery?
Brief Title: Effect of Intranasal Insulin on POCD and POD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hiroaki Sato, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Hiroaki Sato, MD., PhD., Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20184334
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Delirium; Heart Diseases
MeSH Terms: conditions — Delirium; Heart Diseases | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Insulin 40 IU (Experimental): 40 IU of Humulin-R via nose Before surgery and everyday after surgery up to postoperative day 7
  Interventions: Drug: Regular Insulin, Human 100 UNT/ML
- Intranasal Normal Saline (Placebo Comparator): Normal Saline via nose Before surgery and everyday after surgery up to postoperative day 7
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Regular Insulin, Human 100 UNT/ML — 40 IU of Humulin-R to be administered via nose using metered nasal dispenser prior to surgery, and up to 7 days after surgery.
  Other Names: Humulin R
  Arms: Intranasal Insulin 40 IU
Drug: Normal Saline Flush, 0.9% Injectable Solution — Normal Saline to be administered via nose using metered nasal dispenser prior to surgery, and up to 7 days after surgery
  Other Names: Placebo
  Arms: Intranasal Normal Saline

SUMMARY:
Decline in cognitive function after surgery occurs most commonly in older patients and patients undergoing major surgeries, such as heart surgery. Postoperative Cognitive Dysfunction (POCD) may last a prolonged period of time while Postoperative Delirium (POD) is a more acute disturbance in attention, awareness and cognition. The cause of POCD and POD are not fully understood, however some of the pathophysiology of POCD is similar to that of Alzheimer's disease (AD).

Insulin given intravenously during heart surgery has been shown to preserve short and long-term memory function after the operation. Clinical trials further demonstrated that insulin given via the nose (intranasal) improves memory performance of patients with AD or cognitive impairment suggests that intranasal insulin also could be a therapeutic option for POCD and POD.

This study is designed to examine the effect intranasal insulin on POCD and POD. The goal is to investigate whether administration of intranasal insulin during and after heart surgery improves cognitive function postoperatively.

ELIGIBILITY:
Inclusion Criteria:

•elective open heart surgery requiring cardiopulmonary bypass

Exclusion Criteria:

* inability to provide informed consent
* allergy to insulin
* pregnancy
* mother tongue other than English or French
* visual or hearing impairment interfering with the ability to complete cognitive tests.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Confusion Assessment method for the ICU | Up to 7 days after surgery
  Postoperative Delirium is assessment
Rey Auditory Verbal Leaning | up to 12 month
  Episodic Memory Lowest score: 0 Highest Score: 15
Rey-Osterrieth Complex Figure Test | up to 12 month
  Episodic Memory Lowest score: 0 Highest Score: 8

SECONDARY OUTCOMES:
Stroop Test | up to 12 month
  Executive Function
Trail Making Test | up to 12 month
  Executive Function
Tower of London test | up to 12 month
  Executive Function
Symbol Digit Modalities Test | up to 12 month
  Information Processing Speed
Boston Naming Test | up to 12 month
  Language Lowest score: 0 Highest score: 60
Clock Drawing Test | up to 12 month
  Visuospatial Function Lowest score: 1 Highest score: 10

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No